CLINICAL TRIAL: NCT01359462
Title: A Clinical Study of Multiple-dose Pharmacokinetics of Tolvaptan Tablets Administered Orally (15mg Daily) for Consecutively 7 Days in Chinese Patients With Hepatocirrhosis
Brief Title: Multiple-dose Pharmacokinetics Study of Tolvaptan Tablets in Chinese Patients With Hepatocirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Ms. Feng Yan, Otsuka Beijing Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-09-806-01
Record Dates: First submitted 2010-03-05; First posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Hepatic Cirrhosis; Ascites
Keywords: hepatic cirrhosis patients with ascites
MeSH Terms: conditions — Liver Cirrhosis; Ascites | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tolvaptan 15mg tablet (Experimental)
  Interventions: Drug: tolvaptan

INTERVENTIONS:
Drug: tolvaptan — Drug: tolvaptan
  tablet, 15mg, Qd, for 7 days.
  Other Names: SAMSCA

SUMMARY:
For hepatic cirrhosis subjects with ascites or lower extremities, to study Pharmacokinetics, pharmacology, and safety of the drug under fasting condition.

DETAILED DESCRIPTION:
This study is to evaluate the multiple-dose pharmacokinetics, pharmacological actions and safety of Tolvaptan tablets administered orally (15 mg daily) for consecutively 7 days in Chinese adult patients with confirmed Child-Pugh Class B（score 7-9） hepatocirrhosis (accompanied by ascites).

Trial Design:

1. Open, single-center, multi-dose pharmacokinetics study
2. Study population:

   Chinese adult patients with confirmed Child-Pugh Class B (score 7-9) hepatocirrhosis (accompanied by ascites)
3. Dosage and mode of administration of investigational product:

   Oral administration of 1 tablet (15mg) once daily, for consecutive 7 days starting from day 1 of treatment.
4. Study duration:

Screening: 14 days in maximum; Treatment(s): 7 days; Observation: 1 day

ELIGIBILITY:
Inclusion Criteria:

1. Hepatic Cirrhosis with ascites or lower extremities edema
2. Hospitalized patients
3. 18 years old~75 years old
4. Inform Consent Form Signed

Exclusion Criteria:

1. Patients with any of the following diseases, complications or symptoms:

   * Hepatic encephalopathy (coma degree classification note 1 Grade 2 or above);
   * Malignant ascites;
   * Spontaneous bacterial peritonitis;
   * Likely to have gastrointestinal bleeding during the study period;
   * Heart failure (NYHA Note 2 Class Ⅲ andⅣ);
   * Anuria (daily urine output below 100mL);
   * Dysuria induced by urinary tract stenosis, calculus, or tumor.
2. Patients with any of the following history:

   * With gastrointestinal bleeding within 10 days prior to screening;
   * With cerebrovascular accident within 1 month prior to screening;
   * With gout attack within 1 month prior to screening;
   * With allergy or atopy to benzodiazepine drugs (benazepril hydrochloride, etc.).
3. Patients whose systolic blood pressure is below 90mmHg during screening;
4. Patients with abnormal values in the following lab examination indicators:

   Serum creatinine higher than 2.5 times the upper limit of normal range, serum Na+>145mmol/L(or higher than the upper limit of normal range), serum K+> 5.5 mmol/L, uric acid>476µmol/L, child-Pugh score>10
5. Patients ineligible for oral medication
6. Patients in pregnancy or lactation; female of childbearing potential not taking contraceptive measures;
7. Patients having taken blood products including albumin products within 4 days prior to application of investigational product;
8. Patients having participated in clinical trials of other drugs within 1 month prior to screening;
9. Patients used to participate in clinical trials of Tolvaptan and take the said drug;
10. Patients determined by the investigator as illegible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Serum concentration of tolvaptan and its metabolites DM-4103 and DM-4107 | blood sample will be collected at predose, 2,4,6,8,12,24 hour of first drug administration and predose of sixth drug administration and predose,2,4,6,8,12,24 hour of seventh drug administration

SECONDARY OUTCOMES:
pharmacological parameter:Serum concentration of sodium and potassium | Blood sample will be collected at predose on day1;12,24hour of first dosing;before breakfast on day3 to day6;predose and 12,24hour of seventh dosing
pharmacological parameter:24-hr urine | From day-1 to day 8

CONTACTS AND LOCATIONS:
Overall Officials: Minde Zeng, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liu H, Wang Y, Liu T, Chen Y, Zheng X, Liu M, Zhao Q, Zeng M, Jiang J, Mao Y, Hu P. Pharmacokinetics, pharmacodynamics and safety of 15 mg-tolvaptan administered orally for 7 consecutive days to Chinese patients with child-Pugh B cirrhosis. Front Pharmacol. 2024 Jan 26;15:1324299. doi: 10.3389/fphar.2024.1324299. eCollection 2024. PMID 38344178